CLINICAL TRIAL: NCT02695316
Title: Barrier-free Communication in Maternity Care of Allophone Migrants (Barrierefreie Kommunikation in Der Geburtshilflichen Versorgung Allophoner Migrantinnen)
Brief Title: Barrier-free Communication in Maternity Care of Allophone Migrants
Acronym: BRIDGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bern University of Applied Sciences (Other)
Collaborators: Zurich University of Applied Sciences (Other); Swiss Tropical & Public Health Institute (Other); FamilyStart of both Basel (Unknown); Swiss Midwifery Association (Unknown); Federal Office of Public Health, Switzerland (Other Government); Swiss Agency for Combating Racism (Unknown)
Responsible Party: Principal Investigator, Paola Origlia Ikhilor, Prof., Bern University of Applied Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BernUAS
Record Dates: First submitted 2016-02-09; First posted 2016-03-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Expectant and Nursing Mother; Communication; Experiences
Keywords: Migrants; Communication Barriers; Maternal Health Services; Health Services Needs and Demand; Access to Health Care; Professional-Patient Relations; Eritrea; Kosovo; Switzerland
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Migrant Women (Other): Focus Group Discussion in native Language with n=20
  Interventions: Other: Focus Group Discussion in native Language
- Health Care Professionals (Other): Focus Group Discussion with n=20 Health Care Professionals
  Interventions: Other: Focus Group Discussion
- Interpreters (Other): One-to-one Interviews with n=4 intercultural Interpreters
  Interventions: Other: One-to-one Interview
- Telephone Interpreting Protocols (Other): Retrospective quantitative analysis of n=50 Telephone Interpreting Protocols (questionnairs)
  Interventions: Other: Retrospective Quantitative Analysis

INTERVENTIONS:
Other: Focus Group Discussion in native Language — Group Interview with semi-structured key question, moderated in the native language of the participants. Interpreters translate the discussion for the Researcher analogically and adapt it culturally. The discussions are audio-recorded, summarized, translated and transcribed into German.
  Arms: Migrant Women
Other: Focus Group Discussion — Group Interview with semi-structured key question, audio-recorded and ad verbatim transcription
  Arms: Health Care Professionals
Other: One-to-one Interview — One-to-one Interview with semi-structured key question, audio-recorded and ad verbatim transcription.
  Arms: Interpreters
Other: Retrospective Quantitative Analysis — Retrospective Quantitative Analysis of questionnaires (Telephone Interpreting Protocols)
  Arms: Telephone Interpreting Protocols

SUMMARY:
The aim of this study is to describe access and communication barriers of migrant women who do not speak the local language in the Swiss maternity care service provision from the perspective of users, health care professionals and interpreters.

DETAILED DESCRIPTION:
In Switzerland pregnant migrant women and their families are burdened in multiple ways: pregnancy requires an adjustment process and women have to deal with foreign living conditions, limited communication or the uncertainty of their residence status. An increased maternal and child health morbidity and mortality in migrants is well documented. A poor health outcome seems also to be correlated with a limited access to obstetric and maternity care services for migrants. Nearly 10% of foreigners living in Switzerland for more than one year do not speak any of the official languages. In women native of non-EU27 and -EFTA countries and asylum seekers, these rate is considerably higher.

To improve maternity care services for migrants in Switzerland several measures have been taken in the past, e.g. Hospitals for Equity, promotion of transcultural skills, written multilingual health information and interpreter services in hospitals. The availability of comparable measures in outpatient or home care services is rather an exception. One example is the midwives network "FamilyStart", an outpatient institution that offers a helpline and home visiting services for mothers and thier newborns. It collaborates with the National Telephone Interpreter Service.

It is currently unclear how successfully midwives and other health care professionals communicate with allophone migrants, if they use and benefit from any of the currently available support measures and thus may improve the access of migrant women to maternity care in Switzerland.

The study aims

* to describe the access and communication barriers of allophone women with different migration backgrounds in maternity and obstetric health services from the perspective of users, health care professionals and Interpreters
* to make prioritized recommendations on behalf of the Swiss Midwives Association and other professional associations for improving the quality and access of maternity care Services; the transcultural understanding between professionals and users; and the coordination between the different involved services.

It is an exploratory study in three parts:

1. User perspective: Qualitative assessment of the women's experiences. The participants have different migration backgrounds: representatives of the resident foreign population of Switzerland (from Kosovo or Albania with native language Albanian) and asylum seekers (from Eritrea with native language Tigrinya) will be interviewed.
2. Perspective of professionals: Qualitative assessment of the health care professionals experiences and quantitative analysis of protocols of counseling sessions from midwives who have used the telephone interpreting service during a home visit on behalf of FamilyStart.
3. Perspective of interpreters: Qualitative assessment of experiences of professional Interpreters.

ELIGIBILITY:
Group 1: Inclusion criteria:

* healthy women speaking Albanian or Tigrinja
* mothers of a healthy infant up to one year after birth

Exclusion criteria:

* women speaking fluent German
* women with a serious illness during pregnancy, childbirth and/or postpartum or who's infant was seriously ill or died

Group 2: Inclusion criteria:

* Minimum one year working experience
* Experience with allophone Tigrinya or Albanian speaking women

Group 3: Inclusion criteria:

* Female
* Minimum one year working experience
* having either telephone or face-to-face interpreting Expertise

Group 4: No limitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Experiences of migrant women by focus group discussions | after 6 weeks, up to 12 months
  Qualitative description of experiences made with maternity care services during pregnancy, birth, post partum up to one year after birth

SECONDARY OUTCOMES:
Experiences of health care professionals by focus group discussions | within last five years of their professional experience
  Qualitative description of working experiences in maternity care with allohone migrants
Experiences of Interpreters by one-to-one interview | within last five years of their professional experience
  Qualitative description of working experiences when interpreting for pregnant women or mothers in maternity care services
Quality of telephone interpreting consultations with questionnairs | within 24 hours after the consultation
  Descriptive analysis of protocols of telephone interpreted consultations with information on aim, content, perceived benefits and difficulties

CONTACTS AND LOCATIONS:
Overall Officials: Paola Origlia Ikhilor, MSc, Principal Investigator — Bern University of Applied Sciences
Locations (6):
- Switzerland (6):
  - Zurich Universtiy of Applied Sciences, Winterthur, Zurcih
  - FamilyStart, Basel
  - University Hospital Basel, Basel
  - Swiss Midwifery Association SHV, Bern
  - University Hospital Insel Bern, Bern
  - Swiss Service for Telephone Interpreter (Schweizerischer Telefondolmetschdienst ), Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Merten, S., & Gari, S. (2013). Die reproduktive Gesundheit der Migrationsbevölkerung in der Schweiz und anderen ausgewählten Aufnahmeländern. Eine Zusammenfassung der Literatur 2006-2012. Basel: Swiss Tropical and Public Health Institute.
- [Background] Kurth, E. (2013). FamilyStart beider Basel - ein koordinierter Betreuungsservice für Familien nach der Geburt. hebamme.ch(7/8), 35-37.
- [Background] Saladin, P. (Ed.). (2009). Diversität und Chancengleichheit. Grundlagen für erfolgreiches Handeln im Mikrokosmos der Gesundheitsinstitutionen (3. ed.). Bern: Bundesamtes für Gesundheit BAG in Zusammenarbeit mit H+ Die Spitäler der Schweiz.
- [Background] Hermann, M. (2013). Migrationsgerechte Angebote im Bereich reproduktive Gesundheit und frühe Kindheit in der Schweiz. In E. D. d. I. Schweizerische Eidgenossenschaft (Ed.), Eine Bestandesaufnahme von Projekten, Massnahmen und Arbeitsmethoden: Bundesamt für Gesundheit, Sektion Migration und Gesundheit.
- [Background] Bundesamt für Statistik. (2015). Integration - Indikatoren: Sprache - Personen, die 3,2,1 oder keine Landessprache beherrschen. Retrieved 23.03.2015, from Schweizerische Eidgenossenschaft www.bfs.admin.ch/bfs/portal/de/index/themen/
- [Background] Origlia Ikhilor P., van Goch S., Kurth E., Cignacco E. Stocker Kalberer B., Pehlke-Milde J. 2015 Lancierte Studie soll Kommunikation mit allophonen Migrantinnen erleichtern Hebamme.ch 10:4-8
- [Derived] Origlia Ikhilor P, Hasenberg G, Kurth E, Stocker Kalberer B, Cignacco E, Pehlke-Milde J. Barrier-free communication in maternity care of allophone migrants: BRIDGE study protocol. J Adv Nurs. 2018 Feb;74(2):472-481. doi: 10.1111/jan.13441. Epub 2017 Oct 5. PMID 28833465